CLINICAL TRIAL: NCT05690373
Title: Effects of Probiotics in Immune Response to Influenza Vaccination in Adults
Brief Title: Probiotics and Influenza Vaccination Response
Acronym: VERB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: NIZO Food Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTB2022TN106; 200918 (Other: CRO)
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Vaccine Response
Keywords: vaccine response; seroconversion; antibody
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 2B Colony Forming Unit/ day
  Interventions: Dietary Supplement: Probiotic effect on influenza vaccine response
- Placebo (Placebo Comparator): Equivalent placebo
  Interventions: Dietary Supplement: Probiotic effect on influenza vaccine response

INTERVENTIONS:
Dietary Supplement: Probiotic effect on influenza vaccine response — Seroconversion rate: the percentage of subjects achieving at least a 4-fold increase or an increase from >10 to 40 in Ab titre for seronegative subjects.

SUMMARY:
Assess efficacy of oral ingestion of a probiotic product on immune function in a population of healthy adult men and women in a clinical vaccination study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 16 - 65 y and healthy
* Self-reported regular Dutch eating habits as assessed by questionnaire (3 main meals per day)
* No influenza vaccination in 2022
* Non-smokers
* BMI 18.5-28
* Adherence to habitual diet
* no changes during study period
* Signed informed consent

Exclusion Criteria:

* Recent vaccination
* Acute or chronic illness (e.g., diabetes mellitus)
* Gastrointestinal disorders (e.g., inflammatory bowel disease)
* Acute gastroenteritis in the past 2 months
* Immunodeficiency disorder
* Use of immunosuppressive drugs (e.g. cyclosporine, azathioprine, systemic corticosteroids, antibodies)
* Unexplained weight loss or weight gain of > 3 kg in the 3 months prior to pre-study screening
* Alcohol or drug abuse
* Mental status that is incompatible with the proper conduct of the study
* History of cancer
* Use of immune boosting supplements within 4 weeks before screening To be extended & specified in protocol phase

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | From baseline to week 6
  Percentage of subjects achieving at least a 4-fold increase or an increase from >10 to 40 in Antibody titer for seronegative subjects

SECONDARY OUTCOMES:
Change in plasma cytokine levels | Baseline, week 2 and week 6
  Change in plasma cytokine levels (IL-10, IL-4, TFN alpha, IFN gamma)
Change in IgA antibodies against influenza | baseline, week 2, week 6
  Titer of plasma anti-influenza IgA
Change in IgG antibodies against influenza | baseline, week 2, week 6
  Titer of plasma anti-influenza IgG
Change in IgM antibodies against influenza | baseline, week 2, week 6
  Titer of plasma anti-influenza IgM
Change in Gastrointestinal symptoms | baseline, week 2, week 6
  Gastrointestinal manifestations documented through Gastrointestinal Symptom Rating Scale (GSRS, 7-point graded Likert-type scale and includes 15 items combined into 5 symptom clusters - 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms)
Change in Incidence of respiratory infections | baseline, week 2, week 6
  Assessment of respiratory infection through questionnaire (4-point graded Likert-type scale and includes 11 items, including the 8 items comprising the Jackson common cold questionnaire - 0 = absent, 1 = mild, 2 = moderate, 3 = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Alwine Kardinaal, PhD, Study Chair — NIZO food research B.V
Locations (1):
- Alwine Kardinaal, PhD NIZO food research B.V, Ede, Netherlands

IPD SHARING:
Plan to Share IPD: No